CLINICAL TRIAL: NCT03610295
Title: A Novel Prophylactic Peripheral Iridectomy Prevents Aphakic Angle-closure Glaucoma After Congenital Cataract Surgery
Brief Title: Prophylactic Peripheral Iridectomy Prevents Aphakic Angle-closure Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhi Liu, Clinical Professor,director of Zhongshan Ophthalmic Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018KYPJ091
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Congenital Cataract; Aphakic Glaucoma
Keywords: congenital cataract; prophylactic peripheral iridectomy; aphakic angle-closure glaucoma; aphakic open-angle glaucoma; iris posterior synechia; visual axis opacity
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Retrospective,consecutive,nonrandomized comparative trial with historical control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPI group (Experimental): cataract extraction surgery with prophylactic peripheral iridectomy
  Interventions: Procedure: PPI group
- historical control group (Active Comparator): cataract extraction surgery
  Interventions: Procedure: cataract extraction

INTERVENTIONS:
Procedure: PPI group — The patients underwent cataract extraction, posterior capsulotomy, anterior vitrectomy combined with prophylactic peripheral iridectomy.
  Arms: PPI group
Procedure: cataract extraction — The patients underwent cataract extraction, posterior capsulotomy combined with anterior vitrectomy and leave the iris intact.
  Arms: historical control group

SUMMARY:
This is a retrospective, nonrandomized comparative trial with historical control to investigate the safety and efficacy of a novel progressive grasping peripheral iridectomy (PGPI) surgical method in preventing aphakic angle-closure glaucoma (AACG) following congenital cataract surgery.

DETAILED DESCRIPTION:
Aphakic angle-closure glaucoma (AACG) following congenital cataract surgery is a common and serious complication which can be prevented by prophylactic peripheral iridectomy (PPI). However, it is difficult to perform routine PPI via scleral tunnel incision especially when the pupil is dilated. Here, the investigators designed a novel progressive grasping peripheral iridectomy (PGPI) surgical method which can ensure the accurate iridectomy position and minimize the complication. The aim of this study is to assess the safety and efficacy of the PGPI in preventing AACG following congenital cataract surgery.

This is a retrospective, nonrandomized comparative trial with historical control. The congenital cataract patients performed with cataract extraction combined with PPI (PPI group) and the patients performed with cataract extraction alone and leaving the iris intact (historical control group) were enrolled and a retrospective medical chart review was conducted. The IOP, anterior chamber depth, corneal clarity, patency of peripheral iridectomy opening, and the rate of AACG, iris posterior synechia (IPS) and visual axis opacity (VAO) were compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. patients less than 2 years old;
2. patients performed with congenital cataract surgery with or without PPI;
3. patients with routine follow-up at ZOC.

Exclusion Criteria:

1. patients with IOP ≥21 mm Hg or with congenital glaucoma or with a family history of glaucoma;
2. patients with keratopathy, retinopathy, ocular trauma, radiation therapy or intraocular surgery;
3. patients associated with other congenital ocular anomalies, such as anterior segment dysgenesis, microcornea/microphthalmia, persistent fetal vasculature, lens dislocation and iridocoloboma;
4. patients with systemic diseases, such as Down's syndrome, Lowe syndrome, Stickler syndrome, maternal rubella syndrome or trisomy 13.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
The rate of aphakic angle-closure glaucoma | 18-49 months
  Pupillary block with subsequent closure of the filtration angle is the cause of early aphakic angle-closure glaucoma (AACG), which usually happens in the early postoperative period, generally within the first 6 months. AACG presents with elevated IOP (repeatedly >25 mmHg), corneal edema, iris bombe, shallow anterior chamber, peripheral anterior synechia and angle closure.

SECONDARY OUTCOMES:
The rate of iris posterior synechia | 18-49 months
  Postoperative uveal inflammation can result in iris posterior synechia (IPS), referring to the synechia between iris and capsule around pupil. IPS is graded according to the range of the synechia. Grade 0: no synechia; Grade I: <1 quadrant; Grade II: ≤2 quadrants and >1 quadrant ; Grade III: ≤3 quadrants and >2 quadrants; Grade IV: >3 quadrants.
The rate of visual axis opacity | 18-49 months
  visual axis opacification (VAO) refers to developing reopacification of the visual axis in the form of lens proliferation into the visual axis or pupillary membrane.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (2):
- China (2):
  - State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yet-san University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No